CLINICAL TRIAL: NCT06792669
Title: Psychological Assessment and Skills Training by Simulation in Neurosurgery
Acronym: PASSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20150317
Record Dates: First submitted 2015-03-17; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: 300 Students of University of Milan School of Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Neurosimulation training (Experimental): Psychological tests will be administered to the participants aiming at analyzing the psychological profile, the visual-spatial skills, and the manual skills of the medical students. 60 students (under the 10% and over 90% at the tests) - out of a total of 300 students recruited - will be asked to perform 2 medical-surgical tasks (performing an apple debulking by means of a surgical ultrasonic aspirator at the operative microscope and a lumbar puncture on a dedicated manikin); performances will be recorded and rated by experts surgeons. Participants will then perform a microsurgery-training program, by means of specific neurosurgical simulators (Immersive Touch and NeuroTouch) for a defined period of time. Their performances will be recorded and rated by the simulators automatically. After the end of the simulation training program, students will repeat the tasks at the operative microscope and at lumbar puncture manikin, in order to evaluate and quantify their manual skill improvement
  Interventions: Other: Simulation training to evaluate the participants' manual skill improvement

INTERVENTIONS:
Other: Simulation training to evaluate the participants' manual skill improvement

SUMMARY:
The subject of Safety in Health is assuming in time a predominant position with those of high social, economic and political relevance. Numerous medical-surgical procedures are frequently learned as they are performed directly on the patient. The scope of our research, hence, is to recruit 5th- and 6th-year students of Medicine of the University of Milan who will have the opportunity to use two state-of-the-art 3-D virtual reality neurosurgical simulators at the Besta NeuroSim Center. Psychological Evaluation instruments will be used in order to select the personality profile most fit for a career in neurosurgery and to understand what training method is the most appropriate to achieve the best results in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* 5th - 6th year medical students.
* Signed informed consent.

Exclusion Criteria:

• Medical students with any previous surgical experience or simulation training (mechanical, PC-based and/or others).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Simulation training | 4 weeks
  Changes in performances at surgical tasks after a simulation training

SECONDARY OUTCOMES:
Psychological assessment | 4 weeks
  Correlation between cognitive and psycho-attitudinal test and improvement at manual/surgical tasks
Spatial assessment | 4 weeks
  Correlation between tests' results for the visual-spatial ability assessment and the best performances at manual-surgical tasks
Career path | up to 3 years
  Correlation between performances at real/simulated tasks and students' education/career path

CONTACTS AND LOCATIONS:
Overall Officials: Francesco DiMeco, MD, Study Chair — Fondazione Irccs Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto neurologico Carlo Besta, Milan, Milan, Italy